CLINICAL TRIAL: NCT00005793
Title: A Phase I/II Study of Induction Chemotherapy With Daunorubicin, Cytarabine, Topotecan and Etoposide (DATE) for De Novo AML: In the Treatment of Young Patients Ages 16-59
Brief Title: A Phase I/II Study of Induction Chemotherapy With Daunorubicin, Cytarabine, Topotecan and Etoposide
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); SmithKline Beecham (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-11941; CA 82533 (Other: NCI)
Record Dates: First submitted 2000-06-02; First posted 2003-05-07 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Leukemia
Keywords: untreated adult acute myeloid leukemia; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute megakaryoblastic leukemia (M7); adult acute monocytic leukemia (M5b); adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Leukemia, Erythroblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Megakaryoblastic, Acute; Congenital Abnormalities | interventions — Cytarabine; Daunorubicin; Etoposide; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combination Chemotherapy (Experimental): Patients receive induction chemotherapy with daunorubicin IV over 10-15 minutes on days 1-3, cytarabine IV continuously on days 1-5, topotecan IV continuously on days 6-8, and etoposide IV over 60 minutes on days 9 and 10. Within 4 weeks of hematologic recovery, patients achieving remission after induction receive consolidation chemotherapy with cytarabine IV over 1 hour every 12 hours on days 1, 3, and 5. Subsequent courses of consolidation chemotherapy begin within 2 weeks of documentation of hematologic recovery from the prior consolidation course. Consolidation chemotherapy continues for 4 courses in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: Cytarabine; Drug: Daunorubicin; Drug: Etoposide; Drug: Topotecan

INTERVENTIONS:
Drug: Cytarabine
Drug: Daunorubicin
  Other Names: daunorubicin hydrochloride
Drug: Etoposide
Drug: Topotecan
  Other Names: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase I/II trial to study the effectiveness of combination chemotherapy in treating patients who have previously untreated acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) of topotecan when combined with daunorubicin, cytarabine, and etoposide in patients with de novo acute myeloid leukemia.
* Determine the efficacy of this regimen at the MTD of topotecan by measuring the complete response rate in this patient population.
* Determine the days of hospitalization and number of infections associated with this regimen in these patients.
* Correlate serum levels of topotecan and etoposide with the expression of topoisomerase I and II in tumor cells and in peripheral blood mononuclear cells (PBMN), as well as with toxicity and response rate in these patients.
* Correlate tumor cell and PBMN expression and activity of topoisomerase I and II with hematological toxicity and clinical response in these patients.
* Correlate levels of activation of STAT signaling proteins with expression of bcl-2 family proteins and response to chemotherapy in these patients.

OUTLINE: This is a dose-escalation study of topotecan (phase I) followed by a response rate-determination (phase II) study.

Patients receive induction chemotherapy with daunorubicin IV over 10-15 minutes on days 1-3, cytarabine IV continuously on days 1-5, topotecan IV continuously on days 6-8, and etoposide IV over 60 minutes on days 9 and 10. Within 4 weeks of hematologic recovery, patients achieving remission after induction receive consolidation chemotherapy with cytarabine IV over 1 hour every 12 hours on days 1, 3, and 5. Subsequent courses of consolidation chemotherapy begin within 2 weeks of documentation of hematologic recovery from the prior consolidation course. Consolidation chemotherapy continues for 4 courses in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of topotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are accrued to receive induction chemotherapy at the recommended phase II dose.

Patients are followed at 1 month, every 2 months for 1 year, every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 3-36 patients (phase I) and then an additional 24-27 patients (phase II) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed, previously untreated acute myeloid leukemia (AML)

  * All FAB types, M0-M7, excluding M3
  * No AML after myelodysplastic syndrome

PATIENT CHARACTERISTICS:

Age:

* 16 to 59

Performance status:

* Eastern Cooperative Oncology Group (ECOG) 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 2 mg/dL
* SGOT/SGPT normal unless due to leukemic disease
* Alkaline phosphatase normal unless due to leukemic disease

Renal:

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* Ejection fraction at least 50% by MUGA
* No myocardial infarction or serious ventricular arrhythmia within the past 6 months

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other prior malignancy within the past 5 years except resected skin cancer
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior topotecan or any other DNA topoisomerase I inhibitor (e.g., irinotecan, aminocamptothecin, or nitrocamptothecin) or etoposide for any prior malignancy

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Ages: 16 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 1999-07; Primary Completion 2006-07 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 2 years
  Determine the maximum tolerated dose (MTD) of topotecan when combined with daunorubicin, cytarabine, and etoposide in patients with de novo acute myeloid leukemia. Cohorts of 3-6 patients receive escalating doses of topotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Hussain I. Saba, MD, PhD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States